CLINICAL TRIAL: NCT01938339
Title: Development of Clinical Assessment Technique Using Multi-radiotracer PET/MR in Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PETMR-Prostate
Record Dates: First submitted 2013-09-02; First posted 2013-09-10 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Prostate Cancer Recurrent; Stage II Prostate Carcinoma; Stage III Prostate Carcinoma
Keywords: prostate cancer; MRI; PET
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET/MR (Experimental): Multi-radiotracer PET/MR will be performed to compare the accuracy of tumor detection in patient with primary prostate cancer
  Interventions: Device: PET/MR

INTERVENTIONS:
Device: PET/MR — Multi-radiotracer PET/MR will be performed in patients with primary and recurrent prostate cancer
  Other Names: Biograph mMR, Siemens Healthcare

SUMMARY:
To development of clinical assessment technique using multi-radiotracer positron emission tomography/magnetic resonance (PET/MR) in prostate cancer

* to establish the optimal imaging technique of PET/MR using multiple radioactive tracers for prostate cancer
* to establish the imaging biomarker using PET/MR for clinical assessment of prostate cancer and early detection of recurrent prostate cancer

DETAILED DESCRIPTION:
To establish the optimal imaging technique of PET/MR using multiple radioactive tracers for prostate cancer

* Recruiting 30 patients with prostate cancer ahead to radical prostatectomy
* PET/MR using 18F-choline with dedicated prostate MRI in all patients
* PET/MR using 18fluoride(F)-fluorodeoxyglucose(FDG)in all patients after 2-7 days
* PET/CT using 18F-FDG in all patient immediate after 18F-FDG PET/MR
* outcome assessment: comparison of scan time, image quality, tumor detection rate, standardized uptake values of lesions
* establishing optimal imaging technique for prostate PET/MR

To establish the imaging biomarker using PET/MR for clinical assessment of prostate cancer

* comparison of findings on PET/MR, MRI and PET/CT with pathological mapping after radical prostatectomy
* outcome assessment: accuracy of PET/MR for localization and staging of prostate cancer compared with MRI only and PET/CT only

To establish the imaging biomarker using PET/MR for early detection of recurrent prostate cancer

* Recruiting 15 patients with recurrent prostate cancer treated by surgery, hormone, or radiation therapy
* Recruiting 15 patients with treated prostate cancer without recurrence
* PET/MR using 18F-choline with dedicated prostate MRI in all patients
* PET/MR using 18F-FDG in all patients after 2-7 days
* PET/CT using 18F-FDG in all patient immediate after 18F-FDG PET/MR
* comparison of findings on PET/MR, MRI, and PET/CT with clinical data in two patient groups with or without recurrent prostate cancer
* outcome assessment: accuracy of PET/MR for early detection and localization of recurrent prostate cancer compared with MRI only and PET/CT only

ELIGIBILITY:
Inclusion Criteria:

* patient with prostate cancer before treatment
* patient with prostate cancer treated
* patient with prostate cancer recurrent

Exclusion Criteria:

* patient with contraindication for MRI
* Patient with severe renal impairment

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-04 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
accuracy of PET/MR predicting localization and staging of prostate cancer | 1 week after radical prostatectomy
  analysis of accuracy of PET/MR predicting localization and staging of prostate cancer by comparison of PET/MR findings with pathological mapping images after radical prostatectomy

SECONDARY OUTCOMES:
accuracy of early detection and localization of recurrent prostate cancer | 1 week after PET/MR imaging
  accuracy of PET/MR for early detection and localization of recurrence by comparison of PET/MR findings with clinical data in two groups of patients with or without recurrent prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Yeon Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea